CLINICAL TRIAL: NCT00277030
Title: Comparative Trial of Two Strategies of RDS Treatment in Newborns With Birth Weight > 1500 Grams
Brief Title: Two Strategies of RDS Treatment in Newborns With Birth Weight > 1500 Grams
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Sociedad Chilena de Pediatría (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOUC022005
Record Dates: First submitted 2006-01-05; First posted 2006-01-13 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2005-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome; Surfactant; Nasal CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Surface-Active Agents

INTERVENTIONS:
Drug: Surfactant
Device: Nasal CPAP

SUMMARY:
The purpose of this study is to compare two different treatment strategies for RDS in preterm infants > 1500 grams and evaluate whether a selective surfactant administration would reduce the need of intubation, mechanical ventilation and surfactant use.

DETAILED DESCRIPTION:
Respiratory Distress Syndrome (RDS) is a frequent respiratory problem of preterm infants and an important cause of morbidity and mortality.

The management of this disease usually includes intubation, surfactant administration and mechanical ventilation in infants less than 1500 grams. However, in patients over this weight, the treatment has not been standardized and depends on the clinical progression of oxygen requirements.

Hypothesis:

- Early CPAP and selective surfactant administration is an effective treatment for RDS in infants >1500 g. This could decrease or avoid intubation and surfactant administration.

Comparison(s):

Early surfactant administration, when the FiO2 ≥ 0.4. compared to selective surfactant administration when the arterial to alveolar oxygen tension ratio (a/APO2) is ≤ 0.21.

ELIGIBILITY:
Inclusion Criteria:

* Birth Weight > 1500 g.
* First day of life.
* Clinical and radiological signs of RDS.
* Oxygen requirement over 30% to reach an oxygen saturation of 88%.
* Parent's consent approved.

Exclusion Criteria:

* Neonatal asphyxia, 5 minute Apgar < 3 or cord pH <7.0.
* Cardiac or respiratory malformation.
* Chromosomal disease.
* Significative pneumothorax.

Ages: 5 Minutes to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110
Dates: Start 2006-01

PRIMARY OUTCOMES:
The need of intubation and surfactant administration.

SECONDARY OUTCOMES:
Mechanical ventilation and CPAP duration.
Oxygen therapy.
BPD incidence.
Length of stay.
Enteral feeding tolerance.
Air leak.
NEC, gastric perforation.
Death.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Urzua, MD, Principal Investigator — Pontificia Universidad Católica; Alvaro Gonzalez, MD, Study Director — Pontificia Universidad Católica
Locations (3):
- Chile (3):
  - Servicio de Neonatología, Hospital San José, Santiago, Santiago Metropolitan
  - Servicio de Neonatología, Hospital Sótero del Rio, Santiago, Santiago Metropolitan
  - Unidad de Neonatología, Hospital Clínico Pontificia Universidad Católica, Santiago, Santiago Metropolitan

REFERENCES:
- [Background] Gregory GA, Kitterman JA, Phibbs RH, Tooley WH, Hamilton WK. Treatment of the idiopathic respiratory-distress syndrome with continuous positive airway pressure. N Engl J Med. 1971 Jun 17;284(24):1333-40. doi: 10.1056/NEJM197106172842401. No abstract available. PMID 4930602
- [Background] Saunders RA, Milner AD, Hopkin IE. The effects of continuous positive airway pressure on lung mechanics and lung volumes in the neonate. Biol Neonate. 1976;29(3-4):178-86. doi: 10.1159/000240862. PMID 782570
- [Background] Shaffer TH, Koen PA, Moskowitz GD, Ferguson JD, Delivoria-Papadopoulos M. Positive end expiratory pressure: effects on lung mechanics of premature lambs. Biol Neonate. 1978;34(1-2):1-10. doi: 10.1159/000241098. PMID 359057
- [Background] Lindner W, Vossbeck S, Hummler H, Pohlandt F. Delivery room management of extremely low birth weight infants: spontaneous breathing or intubation? Pediatrics. 1999 May;103(5 Pt 1):961-7. doi: 10.1542/peds.103.5.961. PMID 10224173
- [Background] Fujiwara T, Maeta H, Chida S, Morita T, Watabe Y, Abe T. Artificial surfactant therapy in hyaline-membrane disease. Lancet. 1980 Jan 12;1(8159):55-9. doi: 10.1016/s0140-6736(80)90489-4. PMID 6101413
- [Background] Verder H, Albertsen P, Ebbesen F, Greisen G, Robertson B, Bertelsen A, Agertoft L, Djernes B, Nathan E, Reinholdt J. Nasal continuous positive airway pressure and early surfactant therapy for respiratory distress syndrome in newborns of less than 30 weeks' gestation. Pediatrics. 1999 Feb;103(2):E24. doi: 10.1542/peds.103.2.e24. PMID 9925870
- [Background] Avery ME, Tooley WH, Keller JB, Hurd SS, Bryan MH, Cotton RB, Epstein MF, Fitzhardinge PM, Hansen CB, Hansen TN, et al. Is chronic lung disease in low birth weight infants preventable? A survey of eight centers. Pediatrics. 1987 Jan;79(1):26-30. PMID 3797169
- [Background] Gerard P, Fox WW, Outerbridge EW, Beaudry PH. Early versus late introduction of continuous negative pressure in the management of the idiopathic respiratory distress syndrome. J Pediatr. 1975 Oct;87(4):591-5. doi: 10.1016/s0022-3476(75)80832-8. PMID 1099184
- [Background] Krouskop RW, Brown EG, Sweet AY. The early use of continuous positive airway pressure in the treatment of idiopathic respiratory distress syndrome. J Pediatr. 1975 Aug;87(2):263-7. doi: 10.1016/s0022-3476(75)80599-3. PMID 1097619
- [Background] Hegyi T, Hiatt IM. The effect of continuous positive airway pressure on the course of respiratory distress syndrome: the benefits on early initiation. Crit Care Med. 1981 Jan;9(1):38-41. doi: 10.1097/00003246-198101000-00009. PMID 6780266
- [Background] Kamper J, Wulff K, Larsen C, Lindequist S. Early treatment with nasal continuous positive airway pressure in very low-birth-weight infants. Acta Paediatr. 1993 Feb;82(2):193-7. doi: 10.1111/j.1651-2227.1993.tb12637.x. PMID 8477167
- [Background] Lundstrom KE. Initial treatment of preterm infants--continuous positive airway pressure or ventilation? Eur J Pediatr. 1996 Aug;155 Suppl 2:S25-9. doi: 10.1007/BF01958077. PMID 8839743
- [Background] Finer NN, Carlo WA, Duara S, Fanaroff AA, Donovan EF, Wright LL, Kandefer S, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Delivery room continuous positive airway pressure/positive end-expiratory pressure in extremely low birth weight infants: a feasibility trial. Pediatrics. 2004 Sep;114(3):651-7. doi: 10.1542/peds.2004-0394. PMID 15342835
- [Background] Verder H, Robertson B, Greisen G, Ebbesen F, Albertsen P, Lundstrom K, Jacobsen T. Surfactant therapy and nasal continuous positive airway pressure for newborns with respiratory distress syndrome. Danish-Swedish Multicenter Study Group. N Engl J Med. 1994 Oct 20;331(16):1051-5. doi: 10.1056/NEJM199410203311603. PMID 8090164
- [Background] Escobedo MB, Gunkel JH, Kennedy KA, Shattuck KE, Sanchez PJ, Seidner S, Hensley G, Cochran CK, Moya F, Morris B, Denson S, Stribley R, Naqvi M, Lasky RE; Texas Neonatal Research Group. Early surfactant for neonates with mild to moderate respiratory distress syndrome: a multicenter, randomized trial. J Pediatr. 2004 Jun;144(6):804-8. doi: 10.1016/j.jpeds.2004.03.024. PMID 15192630
- [Background] Bernstein G, Mannino FL, Heldt GP, Callahan JD, Bull DH, Sola A, Ariagno RL, Hoffman GL, Frantz ID 3rd, Troche BI, Roberts JL, Dela Cruz TV, Costa E. Randomized multicenter trial comparing synchronized and conventional intermittent mandatory ventilation in neonates. J Pediatr. 1996 Apr;128(4):453-63. doi: 10.1016/s0022-3476(96)70354-2. PMID 8618177
- [Background] Early versus delayed neonatal administration of a synthetic surfactant--the judgment of OSIRIS. The OSIRIS Collaborative Group (open study of infants at high risk of or with respiratory insufficiency--the role of surfactant. Lancet. 1992 Dec 5;340(8832):1363-9. PMID 1360087
- [Background] Stevens TP, Blennow M, Soll RF. Early surfactant administration with brief ventilation vs selective surfactant and continued mechanical ventilation for preterm infants with or at risk for respiratory distress syndrome. Cochrane Database Syst Rev. 2004;(3):CD003063. doi: 10.1002/14651858.CD003063.pub2. PMID 15266470
- [Background] Yost CC, Soll RF. Early versus delayed selective surfactant treatment for neonatal respiratory distress syndrome. Cochrane Database Syst Rev. 2000;(2):CD001456. doi: 10.1002/14651858.CD001456. PMID 10796266